CLINICAL TRIAL: NCT03331575
Title: Hypofractionated vs. Conventionally Fractionated Concurrent CRT for Unresectable Stage III NSCLC
Acronym: HCFCCUSN
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Xiaolong Fu, Xiaolong Fu, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCHLC006
Record Dates: First submitted 2017-10-31; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Unresectable Stage III Non-small-cell Lung Cancer
MeSH Terms: interventions — 26S proteasome non-ATPase regulatory subunit 13

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm1(Hypofractionated Radiotherapy) (Experimental): Hypofractionated Radiotherap（PTV-G60.5Gy/22Fx, 2.75Gy/Fx; PTV-C 49.5Gy/22Fx, 2.25Gy/Fx）, with concurrent chemotherapy : Cisplatin(20 mg/m2 d1) Docetaxel (20 mg/m2 d1),weekly, 6 cycles )
  Interventions: Radiation: Arm1 (Hypofractionated radiotherapy)
- Arms2（Conventional Radiotherapy） (Placebo Comparator): Conventional Radiotherapy（PTV-G60Gy/30Fx,2Gy/Fx; PTV-C 50.4Gy/30Fx, 1.8Gy/Fx）, with concurrent chemotherapy : Cisplatin(20 mg/m2 d1) Docetaxel (20 mg/m2 d1),weekly, 6 cycles )
  Interventions: Radiation: Arm1 (Hypofractionated radiotherapy)

INTERVENTIONS:
Radiation: Arm1 (Hypofractionated radiotherapy) — hypofractionated RT（PTV-G60.5Gy/22Fx, 2.75Gy/Fx; PTV-C 49.5Gy/22Fx, 2.25Gy/Fx）, with concurrent chemotherapy : Cisplatin(20 mg/m2 d1) Docetaxel (20 mg/m2 d1),weekly, 6 cycles )

SUMMARY:
This protocol is a phase III randomized controlled trial (RCT) evaluating the efficacy of hypofractionated vs. conventionally fractionated concurrent chemo-radiotherapy for unresectable stage III non-small-cell lung cancer

DETAILED DESCRIPTION:
Hypofractionated radiotherapy (RT) delivers higher doses of RT over a shorter period of time and may kill more tumor cells and may have fewer side effects. Dose escalation in unresectable stage III NSCLC has been safely achieved up to LEVEL 3 (PTV-G60.5Gy/22Fx, 2.75Gy/Fx; PTV-C 49.5Gy/22Fx, 2.25Gy/Fx). Acute toxicities were well tolerable. Further stage II clinical study has found that hypofractionated RT can significantly improve the efficacy of patients with a low toxicity profile. The aim of this study is to compared with hypofractionated and conventionally fractionated concurrent chemotherapy , and evaluate whether hypofractionated RT can improve local control and overall survival in unresectable stage III non-small-cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 years to 75 years

  •.Histologically proven lung adenocarcinoma or squamous cell lung carcinoma of r Unresectable Stage III NSCLC(according to the TNM classification in theUnion for International Cancer Control (UICC) 7th ed.)
* No prior Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitors (EGFR-TKIs) treatment or other targeted therapy
* No prior thoracic RT
* No severe perioperative complications and expected postoperative lifespan

  ≥4 months
* ECOG Performance Status 0-1
* Voluntarily participated in this study and signed the informed consent form by himself or his agent. Had good compliance with the study procedures, and can cooperate with the relevant examination, treatment and follow-up

Exclusion Criteria:

* Diagnosed with other prior or concurrent malignancies (neoplasm) except for basal cell carcinoma of the skin or carcinoma in situ of the cervix within the last 5 years
* Patients with any severe or uncontrolled systematic disease including severe cardiovascular, liver, kidney, hematopoietic, metabolic disease, or uncontrolled active infection that would preclude study participation
* Patients with positive mental disorder that would preclude study participation;
* Contradictory to chest radiotherapy
* Pregnant or nursing women
* Concurrent other anti-cancer treatment
* Prior Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitors (EGFR-TKIs) treatment or other targeted therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Over survival(OS) | 3years

SECONDARY OUTCOMES:
Disease-free survival (DFS) | 3years

OTHER OUTCOMES:
Locoregional control survival (LCS) | 3years
Distant metastasis-free survival (DMFS) | 3 years
Treatment-related adverse even | 3 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China